CLINICAL TRIAL: NCT00689208
Title: Pharmacological Intervention in Insulin Resistance Targeting Autonomic Nerve Activity - a Concept Study in Mani
Brief Title: Pharmacological Intervention in Insulin Resistance Targeting Autonomic Nerve Activity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Björn Carlsson, MD, PhD, Medical Science Discovery Medicine CDT, AstraZeneca R&D Mölndal, Sweden
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: D4411M00007
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-01

CONDITIONS: Insulin Resistance
Keywords: Clamp
MeSH Terms: conditions — Insulin Resistance | interventions — Atropine; Physostigmine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Atropine — 10 ug/kg bolus, 4 ug/kg/h infusion
Drug: Physostigmine — 0,12ug/kg/min
Drug: Placebo Sodium

SUMMARY:
The present study on pharmacological intervention in autonomic nervous dysregulation(parasympathetic dysfunction,) regarding insulin resistance, is a concept testing in humans tohelp identify potential new pharmacological target sites in the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* BMI of lean and abdominally obese men and women
* weight stable

Exclusion Criteria:

* Ongoing clinically significant diseases
* History of repeated syncope
* resting pulse<50 or systolic blood pressure <100

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Study the effect of anticholinergic drugs on insulin sensitivity by assessment of glucose infusion rate during hyperinsulinemic euglycemic clamp. | After Insulin bolus, following will be measured; p-glucose (every 5 minutes), blood samples (every 30 minutes), pulse (every 5 minutes the first hour then every 10 minutes), blood pressure will be measured (the same as pulse).

SECONDARY OUTCOMES:
Study the effect of cholinergic stimulation on insulin sensitivity by assessment ofglucose infusion rate during hyperinsulinemic euglycemic clamp. | measured; p-glucose (every 5 minutes), blood samples (every 30 minutes), pulse (every 5 minutes the first hour then every 10 minutes), blood pressure will be measured (the same as pulse).
Study the possible difference in effect of cholinergic (physostigmine) andanticholinergic (atropine) drugs on insulin sensitivity in a lean and abdominal obese subgroup of subjects. | measured; p-glucose (every 5 minutes), blood samples (every 30 minutes), pulse (every 5 minutes the first hour then every 10 minutes), blood pressure will be measured (the same as pulse).

CONTACTS AND LOCATIONS:
Overall Officials: Per-Anders Jansson, prof, Principal Investigator — Lundberg Laboratory for diabetic research, Sahlgrenska Universitetssjukhuset Göteborg, Sweden; Jan Eriksson, MSD, Study Chair — Clinical Cardiovascular gastrointestinal departmentAstraZeneca R&D Mölnda Swedenl
Locations (1):
- Research Site, Gothenburg, Sweden